CLINICAL TRIAL: NCT05363618
Title: A Parallel Randomized, Blinded, Un-controlled Tolerability Study of Panosyl-Isomaltooligosaccharides (PIMO) and a Placebo, in Subjects With Heartburn
Brief Title: Tolerability Study of Panosyl-Isomaltooligosaccharides (PIMO) and a Placebo in Subjects With Heartburn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Microbiome Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: MHS-1031-03
Record Dates: First submitted 2022-04-27; First posted 2022-05-06 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Heartburn
Keywords: Heartburn; microbiome; acid reflux; PIMO; indigestion
MeSH Terms: conditions — Heartburn; Gastroesophageal Reflux; Dyspepsia

STUDY DESIGN:
Intervention Model Description: A remote, randomized, blinded, un-controlled trial to evaluate the tolerability of MHS-1031 and separately the tolerability of the formulated placebo in two similar subject groups with heartburn.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Product Tolerability Arm (Active Comparator): Study Product MHS-1031 1g (1.4 ml) per day
  Interventions: Dietary Supplement: Panosyl-isomaltooligosaccharides (PIMO) 1g (1.4 ml)
- Placebo Tolerability Arm (Placebo Comparator): Placebo (Neotame 7.92 mcg/g, phosphoric acid, and sterile water) 1.4 ml per day
  Interventions: Other: Placebo 1.4 ml

INTERVENTIONS:
Dietary Supplement: Panosyl-isomaltooligosaccharides (PIMO) 1g (1.4 ml) — Active study product
  Arms: Product Tolerability Arm
Other: Placebo 1.4 ml — Placebo
  Arms: Placebo Tolerability Arm

SUMMARY:
Remote un-controlled trial to evaluate the tolerability of MHS-1031 and separately the tolerability of the formulated placebo in subjects with heartburn. Candidates will have heartburn and be taking daily PPIs at up to twice the standard OTC or prescription dosage. Approximately 400 subjects (men and women of all races and ethnicities) will be randomly enrolled in a 1:1 ratio to receive Product or Placebo (1.4 ml) per day.

DETAILED DESCRIPTION:
This study will be conducted as a remote un-controlled trial to evaluate the tolerability of MHS-1031 and separately the tolerability of the formulated placebo in two similar subject groups with heartburn. Candidates will have heartburn and be taking daily PPIs at up to twice the standard OTC or prescription dosage.

Approximately 400 subjects (men and women of all races and ethnicities) will be randomly enrolled in a 1:1 ratio to receive Product or Placebo (1.4 ml) per day.

Screening phase: 14 days

Product/Placebo phase: 56 days. From Day 1 through Day 28 each subject will continue taking their usual daily PPI. Beginning on Day 29 and through Day 56 subjects will be requested to not take a PPI. Subjects may re-start taking a PPI at any time.

Product Phase: 28 days. All subjects will receive MHS-1031.

Follow-Up Phase: Subjects who complete the Product Phase of the study will enter into a 14-day Follow-up Phase, during which subjects will take neither placebo nor MHS-1031.

For entry into the Screening Phase, subjects must have the following history: Heartburn experienced at least 1 day per week while taking a PPI.

During the study, tolerability will be assessed via on-line validated PRO questionnaires and assessment of adverse events. Tolerability is defined as no overall worsening of heartburn measurement scores after 8 weeks of taking the product or the placebo compared to baseline scores.

ELIGIBILITY:
Inclusion Criteria:

For Screening Phase inclusion, subjects must meet all the following inclusion criteria to be eligible for enrollment into the study:

1. Subject is willing and able to participate in the study for the required duration, understand and provide signed informed consent, and agrees to undergo all protocol activities.
2. Subject is proficient in reading, writing, and speaking English.
3. Subject is able to complete all required electronic Daily RESQ-eD questionnaires, daily medication questionnaires (Screening Phase, Product/Placebo Phase, Product Phase, and Follow-up Phase), daily General Well-being questionnaire (Screening Phase Only), 4-item Patient Health Questionnaire for Depression and Anxiety (PHQ-4) (Screening Phase Day 14), and monthly Participant Global Assessment questionnaire (Product/Placebo Phase, Product Phase).
4. Have access to a computer/tablet/phone with internet access and active e-mail account in order to complete electronic surveys daily throughout study participation.
5. Males or females between 18 and 75 years of age (inclusive), with a BMI ≥ 19 and < 35 kg/m2.
6. Females must not be pregnant or lactating.
7. Female Subjects of non-childbearing potential whether surgically sterile or postmenopausal
8. Female Subjects of childbearing potential must agree to use adequate contraception from the time of informed consent to the last dose of study product or placebo.
9. Must be on stable doses of medications, if any, prescribed for chronic conditions.
10. Subject must be taking daily PPI (defined as 5 to 7 days per week) of no more than one type (see "a" through "f" below) at no more than twice the standard prescription dose for their specific PPI type, for 4 consecutive weeks prior to the Screening Call, selected from the following list of medications:

    1. omeprazole (no more than 40 mg/day)
    2. esomeprazole (no more than 40 mg/day)
    3. lansoprazole (no more than 60 mg/day)
    4. dexlansoprazole (no more than 60 m/dayg)
    5. pantoprazole (no more than 80 mg/day)
    6. rabeprazole (no more than 40 mg/day)
11. History of a minimum of 3 months of heartburn (ie, "burning feeling behind the breastbone" and/or "pain behind your breastbone" and/or "heartburn" per questions 1, 2 or 3 of RESQ-eD).

Exclusion Criteria:

1. Subject has not maintained a stable diet for ≥ 30 days prior to the Screening Call or is unwilling to maintain a stable diet during the study.
2. Subject has had a surgical procedure requiring general anesthesia < 60 days prior to the Screening Call.
3. Subject has had a colonoscopy in the past 30 days or is scheduled for colonoscopy within the next 4 months and is unable/unwilling to postpone until the completion of study participation.
4. Subject has a history of cancer (other than basal cell carcinoma of the skin) unless the malignancy has been in a complete remission without maintenance therapy (eg, chemotherapy, radiation, surgery) for ≥ 5 years prior to the Screening Call.
5. Subject has any acute or chronic illness that could confound outcome assessments for this study, including, but not limited to:

   1. Known history of untreated peptic or gastric ulcer or Helicobacter pylori (H pylori) positivity without a history of successful treatment.
   2. Known history of ulcerative colitis, Crohn's disease, colon cancer, current stomach ulcers, pancreatitis, diverticulitis
   3. Known history of acute or chronic hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV) infection
   4. Known or suspected alcoholism, drug addiction, or significant drug abuse within 1 year of the Screening Call
6. Subject has any known medical condition, clinical signs and symptoms, vital signs, abnormal laboratory, or other testing, considered clinically significant by the Investigator, that could interfere with the subject's participation in and completion of the study including, but not limited to:

   1. Uncontrolled hypertension
   2. Diabetes uncontrolled by diet (ie, requiring oral medication or insulin)
   3. Previous anaphylactic reaction to any medication
   4. History of adrenal disease, diabetic nephropathy, or gastroparesis
   5. Uncontrolled hypothyroidism
   6. Untreated mental disorder
   7. Spinal cord injury
7. Subject has had a cerebrovascular event (stroke) or myocardial infarction (MI) in the last 6 months
8. Subject has a physiologic or structural abnormality of the GI tract, or disease or condition that can affect GI motility, or defecation
9. Subject has plans to travel outside the USA during the study period
10. Subject has a current COVID19 infection, or a history of a prior COVID19 infection with ongoing symptoms suggestive of "Long COVID"
11. History of scleroderma, Barrett's esophagus, esophageal cancer, esophageal stricture, or esophageal scarring
12. History of endoscopically determined erosive esophagitis of all classes (eg, LA grade A through D)
13. Known hiatal hernia > 2cm
14. History of surgery or endoscopic treatment including fundoplication and dilation for esophageal stricture
15. History of gastric surgery (except for endoscopic removal of benign polyps) or bariatric surgery
16. Subject has had a barium enema within 30 days of the Screening Call
17. Subject has had a fecal impaction that required hospitalization or emergency room treatment within 3 months of the Screening Call
18. Subject has a history diagnosis of an eating disorder in the last 5 years
19. Subject has a history of substantiated (documented by computed tomography (CT) scan or hospitalization) diverticulitis, or any ongoing chronic condition (eg, polycystic kidney disease, endometriosis, ovarian cysts, or other) that may be associated with chronic abdominal pain or discomfort and might confound the assessments in this study during the 2 years prior to the Screening Call
20. Subject has had surgery that meets any of the following criteria:

    1. Gastric bypass surgery or invasive procedure for the treatment of obesity or surgery to remove a segment of the GI tract at any time prior to the Screening Call
    2. Subjects who have had a gastric band unless the band has been completely removed > 60 days prior to the Screening Call
    3. Open surgery of the abdomen, pelvis, or retroperitoneal structures within 6 months prior to the Screening Call
    4. Laparoscopic appendectomy or cholecystectomy or other instrumentation of the bowel < 60 days prior to the Screening Call
21. Prior use of the Study Product MHS-1031
22. History of any the following diseases that can cause heartburn (ie, "burning feeling behind the breastbone" and/or "pain behind your breastbone" and/or "heartburn" per RESQ-eD question 1, 2, or 3): eosinophilic esophagitis, angina, esophageal spasm, achalasia, rumination, or other conditions involving the mouth, throat, dysphagia, or dyspnea
23. Active history of nicotine use, cannabis use, or alcohol abuse (defined as: > 14 drinks/week or 4 drinks/day for men, 7 drinks/week or 3 drinks/day for women). Has used any tobacco, nicotine, or cannabis products (of any type) in the last 6 months or has abused alcohol in the last 6 months
24. Taking any excluded medications listed in the protocol (eg, metformin, antibiotics within the prior 6 months, and during the study)
25. If female, is pregnant, lactating, or intending to become pregnant before or while participating in this study or intending to donate ova during such time period
26. Use of colon prep or high colonic within 30 days prior to the Screening Call
27. Narcotic (eg, opiate) use within 60 days of the Screening Call
28. Antibiotic use within 60 days of the Screening Call
29. Use of any investigational product within 3 months or five half-lives (whichever is longer) prior to study entry
30. Participation in another investigation (clinical trial) during the course of this study
31. Participation in a rigorous weight loss program or have any planned changes in diet or lifestyle, such as getting married, change in residence, change in job, or other highly stressful event
32. Diagnosis of inflammatory bowel disease, irritable bowel syndrome (IBS-D and IBSC), Chronic Idiopathic Constipation
33. Regular use (ie, >=4 times per month) of antibacterial mouthwash (eg, Listerine, Scope, others) and unwilling to stop use for the duration of the study
34. Subject previously took PPIs daily for heartburn, for at least 7 consecutive days in the past, and experienced no improvement
35. Subject is employed by (or is a relative of an employee) or is involved in any way with Microbiome Health Sciences
36. Other conditions or situations that, in the investigator's opinion, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Tolerability as recorded via RESQ-eD (online PRO) questions | 8 weeks
  Tolerability is defined as the proportion of subjects at day 56 with number of days reporting heartburn no greater than baseline. The number of "heartburn days" is defined as the number of days where an answer of >0 (ie, Not "0 - Did not have") is recorded for any of the RESQ-eD questions: "burning feeling behind your breastbone", "pain behind your breastbone", and "heartburn". Subjects who are missing at day 56 will be considered to have not tolerated the study product or to have not tolerated the placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Swann, MD, Principal Investigator — Microbiome Health Sciences
Locations (1):
- Microbiome Health Sciences, Manassas, Virginia, United States

IPD SHARING:
Plan to Share IPD: No